CLINICAL TRIAL: NCT01508390
Title: Phase II Study of Hypofractionated Stereotactic Body Radiation Therapy as a Boost to the Prostate for Treatment of Localized, Non-Metastatic, High Risk Prostate Cancer
Brief Title: Hypofractionated Stereotactic Body Radiation Therapy as a Boost to the Prostate
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-29665
Record Dates: First submitted 2011-12-09; First posted 2012-01-12 (Estimated); Last update posted 2025-06-26 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
Keywords: prostate
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Radiosurgery; Radiation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Boost (Experimental): CyberKnife Boost 21 Gy in 7 Gy per day, 3 fractions, Every other day
  Interventions: Radiation: CyberKnife Boost

INTERVENTIONS:
Radiation: CyberKnife Boost — 21 Gy in 7 Gy per day, 3 fractions, Every other day
  Other Names: stereotactic radiotherapy, cyberknife, radiation

SUMMARY:
In this study, participants will have standard Androgen Deprivation Therapy and undergo standard external beam radiation therapy to the prostate and at-risk lymph nodes by Intensity Modulated Radiation Therapy. The subsequent *boost* radiation therapy to the prostate alone will be given using the CyberKnife, rather than using the standard Intensity Modulated Radiation Therapy. This study will also see how CyberKnife affects the quality of the participant's life.

DETAILED DESCRIPTION:
In this study, participants will have standard androgen deprivation therapy and undergo standard radiation therapy to the prostate and at-risk lymph nodes by intensity-modulated radiation therapy (IMRT). The subsequent *boost* radiation therapy to the prostate alone will be given using the CyberKnife, rather than using the standard Intensity Modulated Radiation Therapy. This study will also see how CyberKnife affects the quality of the participant's life.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically proven adenocarcinoma of the prostate

   1. Gleason score (2-10)
   2. Biopsy within six months of date of registration
   3. Patient age >18 years
2. Clinical stage (American Joint Committee on Cancer 7th Edition)

   a. T-stage determined by physical exam (Digital Rectal Exam Required)

   i. MRI findings (e.g. extracapsular extension) can be used to determine T-staging

   b. N-stage determined using abdominopelvic CT scan and/or MRI

   c. M-stage determined by physical exam, CT and/or MRI, and bone scan (must be M0, excepting Lymph nodes)

   Please note: a SPECT bone scan including a CT of the abdomen and pelvis or an F18 Fluciclovine PET/CT fulfills protocol criteria for both the abdominopelvic CT and bone scan.
3. Patients must belong to one of the following risk groups:

   * PSA > 20 and < 150 and/or
   * Gleason 8-10 and/or
   * > clinical T3a and/or
   * Clinical N1

   OR
   * PSA 10 - 20 AND
   * Gleason 7 AND
   * Clinical T2b - T2c
4. Patient is receiving, or planning to receive standard androgen deprivation therapy and initial IMRT to the prostate and positive or at-risk lymph nodes.
5. Prostate volume greater than 20 cc and less than 100 cc
6. Eastern Cooperative Oncology Group (ECOG) performance status 0-1
7. Patient has agreed to complete questionnaires
8. Signed IRB approved informed consent
9. Patient eligible to have an MRI
10. Must be able to tolerate the confinement of an MRI procedure

Exclusion Criteria:

1. No prior prostate surgery (including TURP) or prostate cancer treatment with the exception of androgen deprivation therapy
2. No prior radiotherapy to the pelvis
3. No implanted hardware (including metal) or other material that would prohibit appropriate treatment planning or treatment delivery
4. No metastatic disease, with the exception of lymph node positive disease
5. No chemotherapy for a malignancy in the last 5 years.
6. No history of an invasive malignancy (other than basal or squamous skin cancers) in the last 5 years.
7. No heart pacemaker, No metallic foreign body (metal sliver) in the eye, No aneurysm clip in the brain
8. No history of a pelvic or horseshoe kidney
9. No diagnosis of inflammatory bowel disease

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2011-06 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Document rate of biochemical Disease-Free Survival (bDFS) | 5 years
  To document the rate of biochemical Disease-Free Survival (bDFS), American Society for Radiation Oncology definitions

SECONDARY OUTCOMES:
Rate of local failure | 5 years
  Rate of local failure
Rate of distant failure | 5 years
  Rate of distant failure
disease-free survival | 5 years
  disease-free survival
Rate of disease-specific survival | 5 years
  Rate of disease-specific survival
Rate of overall survival | 5 years
  Rate of overall survival
Estimate the rates of acute and late grade 3-5 gastrointestinal and genitourinary toxicity | 5 years
  rates of acute and late grade 3-5 gastrointestinal and genitourinary toxicity following combination androgen deprivation therapy, External Beam Radiation Therapy and CyberKnife radiosurgery as a boost

CONTACTS AND LOCATIONS:
Overall Officials: Ariel Hirsch, MD, Principal Investigator — Boston Medical Center
Locations (1):
- Boston Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No